CLINICAL TRIAL: NCT03028831
Title: Randomized Controlled Trial of Resistant Starch to Reduce Colon Cancer Risk in Alaska Native People.
Brief Title: Fiber to Reduce Colon Cancer in Alaska Native People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other)
Responsible Party: Principal Investigator, Stephen O'Keefe, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO16080079
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2022-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: dietary supplementation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: similar packets, similar appearing supplements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch (Active Comparator): 70g high-amylose maize starch which contains 42g of type 2 resistant starch
  Interventions: Dietary Supplement: Resistant starch
- Digestible Starch (Placebo Comparator): 70g of fully digestible starch comprised of amylopectin corn starch.
  Interventions: Dietary Supplement: 70g of fully digestible starch amylopectin corn starch

INTERVENTIONS:
Dietary Supplement: 70g of fully digestible starch amylopectin corn starch — Fully digestible amylopectin corn starch
  Arms: Digestible Starch
Dietary Supplement: Resistant starch — 70g high-amylose maize starch
  Arms: Resistant Starch

SUMMARY:
Alaska native people (AN) have the highest recorded incidence and death rate from colon cancer in the world (>90:100,000). We hypothesize that the AN, despite their high consumption of anti-inflammatory and antineoplastic n-3 fish oils, are at increased risk of colon cancer because of colonic butyrate deficiency resulting from their remarkably low consumption of fiber-containing foods. We hypothesize that fiber supplementation of their usual diet will result in a bloom of butyrate producing microbes in the colon, resulting in increased butyrate production, which will suppress their high microbial secondary bile acid production, antagonize the actions of other food (smoked fish) and environmental carcinogens (tobacco, alcohol), and interact with the high circulating levels of n-3 fish oils to suppress colonic inflammation and cancer risk. In order to investigate this, we will conduct a randomized double-blinded 4-week clinical trial in up to 100 randomizable healthy, middle-aged AN undergoing screening colonoscopy, with the objective of obtaining 60 completed interventions. The interventions will consist of either a high-dose soluble fiber supplement given as a drink, together with their usual diet which currently contains about 15g total fiber/d, or to a control digestible starch drink plus their usual diet. The primary endpoint will be a clinically significant reduction in Ki67 proliferative colonic mucosal biomarkers of cancer risk. Microbiome and metabolome mechanisms responsible for the anticipated changes in mucosal biomarkers will also be investigated. Our results in extreme risk AN will be further evaluated by comparison to similar measurements previously made in minimal risk rural Africans and intermediate risk African Americans. Our results will be used to provide the scientific basis for a definitive large-scale high-fiber supplementation study (to achieve >50g total fiber/d) to suppress adenomatous polyp recurrence following colonoscopy.

DETAILED DESCRIPTION:
Randomization for the double blind, placebo controlled, clinical trial: Recruitment will continue until 60 volunteers have completed the intervention study. Based on previous experience with similar studies, we anticipate 20% of screened patients to be ineligible or drop out, which means, so we plan on consenting and screening approximately 100 potential participants. Baseline data from these participants will be retained. Individuals will be randomized via minimisation (based on age, sex, polypectomy, high fish consumption, and BMI - factors that might influence microbiota composition and function)) to either the resistant starch (RS) group or the control digestible starch (DS) group upon completion of the Stabilization Period.

1. RS Group: Participants will continue with their usual diet plus fiber supplement given as a daily dose of 70g high-amylose maize starch (HAM-RS, HI-MAIZE®260: Ingredion Incorporated, Bridgewater, NJ), which contains 42g of type 2 resistant starch, for 4 weeks. Data from previous studies[69] suggests that their usual diet will contain approximately 13g dietary fiber/day, chiefly insoluble, indicating that total fiber intake would be approx. 55g/d. Supplements will be pre-weighed out in batches from the same source and kept in airtight containers. The supplement may be taken as a single or divided dose dissolved in 250ml water, low fat milk, or orange juice
2. DS (Control) Group participants will continue on their usual diet, plus 70g of fully digestible starch (waxy corn starch comprised of amylopectin, AMIOCA® corn starch, Ingredion Incorporated, Bridgewater, NJ ) weighed out, analyzed, and prepared as previously. The RS and control supplements will appear and taste similar, allowing for coding and distribution in a double-blind fashion. The supplements will be equicaloric.

Interventions will include fecal and colonic content sampling for measurement of the microbiome and metabolome, and flexible sigmoidoscopy to obtain mucosal biopsies before and after the dietary supplementation.

Monitoring During the Clinical Trial: This will follow the scheme laid out on Figure 7. On day 0, participants will visit the clinic and will be asked to save their first fecal sample using our standard operating procedure developed and proven to be effective in our last study. They will then be given their first supplement drink made up in their vehicle of choice, and taken with a standard meal provided by the diet kitchen. During the trial, they will be instructed on the use of a simple diary to be completed at home. This will record the major food items consumed each day, the timing and completion of drink supplements, as well as the bowel function questionnaire to assess daily GI tolerance, i.e. abdominal discomfort, distension, gas, bowel frequency, nausea, vomiting. They will be asked to return to the clinic for a follow-up appointment on day 7, 14 and 21 in order to repeat the fecal and breath tests described above. At the same time, body weight will be monitored using one scale. At the end of 4 weeks, participants will be asked to return to the clinic for repeat of the colonic sampling performed at baseline.

ELIGIBILITY:
Inclusion Criteria: Healthy AN volunteers (from GI standpoint) between 40-70 years (age at which colon cancer screening colonoscopy is recommended in this population) and BMI between 18-40 Kg/m2. It should be noted that in our previous study, we found no difference in the responses of the key parameters (mucosal biomarkers, butyrate and secondary bile acid producers, fecal SCFA and bile acids) to increased fiber diets between those with normal body weight, those overweight, and those who were obese (Nature Comm Supplement). Patients who have, or have had noncancerous polyps removed previously by colonoscopy will be eligible. Alaska Native race will be defined as those eligible to receive health care through the Alaska Tribal Health System. Exclusion criteria: These are detailed under Human Subjects. Participants will be ineligible if they have a history of familial adenomatous polyposis or hereditary non-polyposis colorectal cancer, or have previous colonoscopic evidence of inflammatory bowel disease or colon cancer. Also ineligible will be individuals with known renal, hepatic, or bleeding disorders; previous GI surgery resulting in disturbed gut function due to of loss of bowel or altered anatomy; or any form of chronic GI disease resulting in disturbed gut function, diarrhea, and malabsorption. Individuals with antibiotic use within the past 12 weeks, current steroids use, or on medical treatment for diabetes, will also be excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
colonic mucosal proliferation | 4 weeks
  biomarker of cancer risk

SECONDARY OUTCOMES:
colonic microbiota | 4 weeks
  fecal and colonic microbiota analysis
colonic secondary bile acids | 4 weeks
  fecal and colonic conjugated bile acid analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Riscuta, Study Director — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Alaskan Native Tribal Health Consortium, Anchorage, Alaska
  - Upittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
we will use a public deposit when all the data analysis is completed
Time Frame: 2012
Access Criteria: public

REFERENCES:
- [Background] O'Keefe SJ. Diet, microorganisms and their metabolites, and colon cancer. Nat Rev Gastroenterol Hepatol. 2016 Dec;13(12):691-706. doi: 10.1038/nrgastro.2016.165. Epub 2016 Nov 16. PMID 27848961
- [Result] O'Keefe SJ, Li JV, Lahti L, Ou J, Carbonero F, Mohammed K, Posma JM, Kinross J, Wahl E, Ruder E, Vipperla K, Naidoo V, Mtshali L, Tims S, Puylaert PG, DeLany J, Krasinskas A, Benefiel AC, Kaseb HO, Newton K, Nicholson JK, de Vos WM, Gaskins HR, Zoetendal EG. Fat, fibre and cancer risk in African Americans and rural Africans. Nat Commun. 2015 Apr 28;6:6342. doi: 10.1038/ncomms7342. PMID 25919227
- [Result] Ou J, Carbonero F, Zoetendal EG, DeLany JP, Wang M, Newton K, Gaskins HR, O'Keefe SJ. Diet, microbiota, and microbial metabolites in colon cancer risk in rural Africans and African Americans. Am J Clin Nutr. 2013 Jul;98(1):111-20. doi: 10.3945/ajcn.112.056689. Epub 2013 May 29. PMID 23719549
- [Result] Koller KR, Wilson A, Normolle DP, Nicholson JK, Li JV, Kinross J, Lee FR, Flanagan CA, Merculieff ZT, Iyer P, Lammers DL, Thomas TK, O'Keefe SJD. Dietary fibre to reduce colon cancer risk in Alaska Native people: the Alaska FIRST randomised clinical trial protocol. BMJ Open. 2021 Aug 27;11(8):e047162. doi: 10.1136/bmjopen-2020-047162. PMID 34452959